CLINICAL TRIAL: NCT00789906
Title: Development of Population Norms of the Computerized Neuropsychological Assessment for Effectiveness of the Antipsychotic Treatment in Schizophrenia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: BeerYaakov Mental Health Center (Other Government)
Responsible Party: Semion Kertzman, BeerYaakov Mental Health Center
Other Study IDs: 223CTIL
Record Dates: First submitted 2008-11-11; First posted 2008-11-13 (Estimated); Last update posted 2008-11-13 (Estimated); Status verified 2008-11

CONDITIONS: Schizophrenia
Keywords: Computerized Neuropsychological Assessment; Development of Population Norms of the Computerized Neuropsychological Assessment
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- 1: 350 healthy women , aged from 18 to 89
- 2: 350 healthy men, aged from 18 to 89

SUMMARY:
Schizophrenia affects cognition, emotion, and behavior. Neuropsychological assessment enables a better understanding of antipsychotic effectiveness and the brain processes, underlying cognitive functioning in schizophrenia.

Neurocognitive deficits in schizophrenia patients appears to explain up to 61% of the variance of functional outcome and is an important predictor of social reintegration (Peuskens et al, 2005) and independent living activitiy (Green et al, 2004). Impaired social functioning within schizophrenia population has been associated with increased health-care costs. Since social and occupational disability may generate the largest indirect costs of the illness, treatment of cognitive deficits has an enormous impact on the cost and disability associated with schizophrenia (McGurk and Mueser, 2004).

However, the gap between cognitive science and clinical practice limits the implementation of cognitive assessment in the routine evaluation of schizophrenia patients. Pharmaceutical industry initiated numerous large scale, multisite studies on the impact of novel antipsychotics on cognitive deficits in schizophrenia patients.

The aim of this research is to develop population norms of the computerized neuropsychological assessment for effectiveness of the antipsychotic treatment in schizophrenia.

ELIGIBILITY:
Inclusion Criteria:

* An IQ, which is within normal range.

Exclusion Criteria:

* Psychiatric co-morbidity.
* Physical disability or illness.
* A history of severe head injury.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 700 healthy adults (350 women and 350 men, aged from 18 to 89)
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2008-07

CONTACTS AND LOCATIONS:
Locations (1):
- Beer-Yaacov MHC, Beer Yaacov, Israel